CLINICAL TRIAL: NCT02583074
Title: Subthalamic Deep Brain Stimulation in Patients With Medication-Refractory Primary Cranial-Cervical Dystonia: A Randomised, Sham-controlled Trial
Brief Title: Clinical Trial of STN-DBS for Primary Cranial-Cervical Dystonia
Acronym: STN-CCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Kai Zhang, PhD，MD, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZYLX201305
Record Dates: First submitted 2015-09-23; First posted 2015-10-21 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Dystonia
Keywords: deep brain stimulation; Subthalamic Nucleus; dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation Group (Experimental): Patients in 'Neurostimulation Group' will receive subthalamic nucleus deep brain stimulation for 3 months.
  Interventions: Procedure: Stimulation
- Sham-stimulation Group (Sham Comparator): Patients in 'Sham-stimulation Group' will receive sham stimulation of subthalamic nucleus for 3 months.
  Interventions: Procedure: Sham-stimulation

INTERVENTIONS:
Procedure: Stimulation — After surgery, patients in 'Neurostimulation Group' will receive subthalamic nucleus stimulation for 3 months.
  Arms: Stimulation Group
Procedure: Sham-stimulation — After surgery, patients in 'sham-stimulation Group' will receive subthalamic nucleus sham-stimulation for 3 months.
  Arms: Sham-stimulation Group

SUMMARY:
Primary cranial-cervical dystonia is managed mainly by repeated botulinum toxin injections.This study is to establish whether subthalamic nucleus neurostimulation could improve symptoms in patients not adequately responding to chemodenervation or oral drug treatment. Investigators compared this surgical treatment with sham stimulation in a randomized, controlled clinical trial.

DETAILED DESCRIPTION:
In this randomised, sham-controlled trial, investigators will recruit forty patients with primary cranial-cervical dystonia to receive an implanted device for STN-DBS, and participants will be randomly assigned to receive either neurostimulation or sham stimulation for 3 months.The primary end point was the change from baseline to 3 months in the severity of symptoms, according to the Burke-Fahn-Marsden Dystonia Rating Scale. Two masked dystonia experts who unaware of treatment status will assess the severity of dystonia by reviewing standardised videos.Subsequently, all patients will receive open-label neurostimulation; blinded assessment will be repeated after 6 months of active treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of primary cranial-cervical dystonia: blepharospasm combined with dystonia of the lower facial muscles. Cervical muscles can be involved but did not dominate the clinical picture.
2. Medical intractable：including various drugs and local botulinum toxin injections.
3. patients deteriorated in activities of daily living and showed social withdrawal during the course of their disease as they suffered from apparent hyperkinesia of facial muscles and functional blindness secondary to severe blepharospasm.

Exclusion Criteria:

1. All other topographical areas remained unaffected.
2. Secondary causes will be excluded by standard cranial magnetic resonance imaging (MRI) scans.
3. Cognitive impairment, dementia,severe psychiatric diseases as well as higher surgical risks due to comorbidities will also be exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09-15; Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of motor and disability scores | Baseline,3 months after surgery, 6 months after active stimulation
  Burke-Fahn-Marsden Dystonia Rating Scale (movement and disability scores, BFMDRSM/D)

SECONDARY OUTCOMES:
Quality of life | Baseline,3 months after surgery,6 months after active stimulation
  SF-36
Depression | Baseline,3 months after surgery,6 months after active stimulation
  Beck Depression Inventory

OTHER OUTCOMES:
Adverse event | 3 months after surgery,6 months after active stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Jian-guo, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing

REFERENCES:
- [Result] Skogseid IM. Pallidal deep brain stimulation is effective, and improves quality of life in primary segmental and generalized dystonia. Acta Neurol Scand Suppl. 2008;188:51-5. doi: 10.1111/j.1600-0404.2008.01032.x. PMID 18439222
- [Result] Limotai N, Go C, Oyama G, Hwynn N, Zesiewicz T, Foote K, Bhidayasiri R, Malaty I, Zeilman P, Rodriguez R, Okun MS. Mixed results for GPi-DBS in the treatment of cranio-facial and cranio-cervical dystonia symptoms. J Neurol. 2011 Nov;258(11):2069-74. doi: 10.1007/s00415-011-6075-0. Epub 2011 May 7. PMID 21553081
- [Result] Reese R, Gruber D, Schoenecker T, Bazner H, Blahak C, Capelle HH, Falk D, Herzog J, Pinsker MO, Schneider GH, Schrader C, Deuschl G, Mehdorn HM, Kupsch A, Volkmann J, Krauss JK. Long-term clinical outcome in meige syndrome treated with internal pallidum deep brain stimulation. Mov Disord. 2011 Mar;26(4):691-8. doi: 10.1002/mds.23549. Epub 2011 Feb 10. PMID 21312284
- [Result] Ostrem JL, Markun LC, Glass GA, Racine CA, Volz MM, Heath SL, de Hemptinne C, Starr PA. Effect of frequency on subthalamic nucleus deep brain stimulation in primary dystonia. Parkinsonism Relat Disord. 2014 Apr;20(4):432-8. doi: 10.1016/j.parkreldis.2013.12.012. Epub 2014 Jan 5. PMID 24440061
- [Result] Cao C, Pan Y, Li D, Zhan S, Zhang J, Sun B. Subthalamus deep brain stimulation for primary dystonia patients: a long-term follow-up study. Mov Disord. 2013 Nov;28(13):1877-82. doi: 10.1002/mds.25586. Epub 2013 Jul 16. PMID 23861342